CLINICAL TRIAL: NCT03684616
Title: Epidemiology, Management, Prognosis and Medical Cost Analysis of In-hospital and Out-of-hospital Cardiac Arrest Patients
Brief Title: Epidemiology, Management, Prognosis and Medical Cost Analysis of IHCA and OHCA
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201404063W; NHRI database (Registry Identifier: National Taiwan University Hospital)
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2014-05

CONDITIONS: Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Statin treatment prior to cardiac arrest
  Interventions: Drug: Statin
- No Statin treatment prior to cardiac arrest
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: Statin — continuous statin treatment for 3 months prior to cardiac arrest

SUMMARY:
The study is a retrospective analysis of Taiwan national health insurance in cardiac arrest patients. The factors related to the outcomes of cardiac arrest patients were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* out-of-hospital cardiac arrest,

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The out-of-hospital cardiac arrest patients from 2004-2012 were included for analysis
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2014-05-08 (Actual); Primary Completion 2015-05-07 (Actual); Study Completion 2015-05-07 (Actual)

PRIMARY OUTCOMES:
one year survival | up to one year

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No